CLINICAL TRIAL: NCT00837213
Title: Comparative Efficacy and Safety of Benzoyl Peroxide Used in Combination With Clindamycin vs. Benzoyl Peroxide Used in Combination With Clindamycin and Doxycycline in the Treatment of Moderate Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EVF0701
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Results first posted 2010-08-31 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Acne
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Benzoyl Peroxide; Clindamycin; Acne RA-1,2; Doxycycline

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BPO with clindamycin foam (Active Comparator): Benzoyl peroxide (BPO) wash with clindamycin foam
  Interventions: Drug: Benzoyl peroxide with clindamycin
- BPO + clindamycin foam + doxycycline (Active Comparator): Benzoyl peroxide (BPO) wash with clindamycin foam and doxycycline capsules
  Interventions: Drug: Benzoyl peroxide with clindamycin and doxycycline

INTERVENTIONS:
Drug: Benzoyl peroxide with clindamycin — Benzoyl peroxide wash - Clindamycin foam
  Other Names: Acne
  Arms: BPO with clindamycin foam
Drug: Benzoyl peroxide with clindamycin and doxycycline — Benzoyl peroxide wash - Clindamycin foam - Doxycycline capsules
  Other Names: Acne
  Arms: BPO + clindamycin foam + doxycycline

SUMMARY:
To compare the efficacy and safety of Benzoyl peroxide used in combination with clindamycin vs. Benzoyl peroxide used in combination with clindamycin and doxycycline in the treatment of moderate acne

DETAILED DESCRIPTION:
To compare the efficacy and safety of Benzoyl peroxide used in combination with clindamycin vs. Benzoyl peroxide used in combination with clindamycin and doxycycline once daily in the treatment of moderate acne

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with acne vulgaris . Able to understand the requirements of the study and sign informed consent/HIPAA authorization forms.

Exclusion Criteria:

* Known hypersensitivity to any of the components of the study drugs or used of prohibited medications or any medical condition that contraindicate the subject's participation in the clinical study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - Center for Dermatology, Cosmetic and Laser Surgery, Fremont, California
  - Las Vegas Skin & Cancer Clinic, Las Vegas, Nevada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: First Subject Enrolled May 2008, Last Subject completed August 28, 2008.
  Types of location: Dermatology Research Center
Groups:
- Benzoyl Peroxide Wash -Clindamycin Foam: Benzoyl peroxide wash applied in the shower or bath daily with Clindamycin foam applied after the shower or bath daily.
- Benzoyl Peroxide Wash -Clindamycin Foam -Doxycycline Capsules: Benzoyl peroxide wash applied in the shower or bath daily with Clindamycin foam applied after the shower or bath daily. Doxycycline 100 mg capsules were taken once a day.
Period: Overall Study
Arm/Group | Benzoyl Peroxide Wash -Clindamycin Foam | Benzoyl Peroxide Wash -Clindamycin Foam -Doxycycline Capsules
Started | 16 | 17
Completed | 10 | 12
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — not stated | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benzoyl Peroxide Wash -Clindamycin Foam | Benzoyl Peroxide Wash -Clindamycin Foam -Doxycycline Capsules | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.9 (8.5) | 21.9 (6.9) | 22.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 9 | 8 | 17
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 10 | 12 | 22
  Asian | 3 | 0 | 3
  Hispanic | 2 | 3 | 5
  Black or African American | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Inflammatory Acne Lesions From Baseline to Week 16
Description: Percent change from baseline to week 16 in inflammatory acne lesions (pustules/papules)(chest and back)
Time Frame: Baseline, Week 16
Population: ITT
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Benzoyl Peroxide Wash -Clindamycin Foam | Benzoyl Peroxide Wash -Clindamycin Foam -Doxycycline Capsules
Number analyzed (Participants) | 16 | 17
Percent change | -52.70 (26.83) | -48.84 (40.37)

2. Primary Outcome: Percent (%) Change in Non-inflammatory Acne Lesions From Baseline to Week 16.
Description: Percent change in Non-inflammatory acne lesions (whiteheads and blackheads)(chest and back) from baseline to week 16.
Time Frame: Baseline, Week 16
Population: ITT
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Benzoyl Peroxide Wash -Clindamycin Foam | Benzoyl Peroxide Wash -Clindamycin Foam -Doxycycline Capsules
Number analyzed (Participants) | 16 | 17
Percent Change | -25.27 (45.64) | -44.69 (43.72)

3. Primary Outcome: Percent Change in Total Acne Lesion Counts From Baseline to Week 16
Description: Percent change from baseline to week 16 in total acne lesions (inflammatory + non-inflammatory)
Time Frame: Baseline, Week 16
Population: ITT
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Benzoyl Peroxide Wash -Clindamycin Foam | Benzoyl Peroxide Wash -Clindamycin Foam -Doxycycline Capsules
Number analyzed (Participants) | 16 | 17
Percent Change | -38.49 (33.06) | -46.11 (39.74)

4. Secondary Outcome: Percent (%) Change in Inflammatory Lesion Counts (Chest and Back) From Baseline to Week 12
Description: Percent change in inflammatory lesion counts (chest and back)from Baseline to Week 12
Time Frame: Baseline, Week 12
Population: ITT
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Benzoyl Peroxide Wash -Clindamycin Foam | Benzoyl Peroxide Wash -Clindamycin Foam -Doxycycline Capsules
Number analyzed (Participants) | 16 | 17
Percent Change | -49.04 (31.63) | -45.44 (46.09)

5. Secondary Outcome: Percent Change in Non-inflammatory Lesions (Chest and Back) From Baseline to Week 12
Description: Percent change in non-inflammatory lesions (chest and back) from baseline to Week 12
Time Frame: Baseline, Week 12
Population: ITT
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Benzoyl Peroxide Wash -Clindamycin Foam | Benzoyl Peroxide Wash -Clindamycin Foam -Doxycycline Capsules
Number analyzed (Participants) | 16 | 17
Percent change | -38.43 (39.75) | -38.52 (39.03)

6. Secondary Outcome: Percent Change in Total Lesions (Chest and Back) From Baseline to Week 12
Description: Percent change in total lesions (chest and back) from baseline to Week 12
Time Frame: Week 12
Population: ITT
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Benzoyl Peroxide Wash -Clindamycin Foam | Benzoyl Peroxide Wash -Clindamycin Foam -Doxycycline Capsules
Number analyzed (Participants) | 16 | 17
Percent change | -44.16 (29.41) | -41.74 (38.56)

7. Primary Outcome: Change in Investigator Global Assessment (IGA)
Description: Change in Investigator Global Assessment (IGA) Average values chest and back.
  IGA scale:
  0 - Clear
  0.5 - Clear/almost clear
  1. Almost Clear
     1.5- Almost Clear/Mild
  2. Mild
     2.5- Mild/Moderate
  3. Moderate
  3.5- Moderate/Severe
Time Frame: Baseline, Weeks 4, 8,12, and 16
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Benzoyl Peroxide Wash -Clindamycin Foam | Benzoyl Peroxide Wash -Clindamycin Foam -Doxycycline Capsules
Number analyzed (Participants) | 16 | 17
Units on a scale
  Change from Baseline to Week 4 | -0.42 (0.57) | -0.61 (0.59)
  Change from Baseline to Week 8 | -0.55 (0.88) | -0.85 (0.72)
  Change from Baseline to Week 12 | -1 (1.07) | -1.09 (0.8)
  Change from Baseline to Week 16 | -0.9 (0.94) | -1.25 (0.97)

8. Secondary Outcome: Percentage of Particpants With IGA Score at Week 16
Description: Investigator Global Assessment (IGA) at Week 16 based on the Investigator Global Assessment
  IGA:
  0 - Clear
  0.5 - Clear/almost clear
  1. Almost Clear
     1.5- Almost Clear/Mild
  2. Mild
     2.5- Mild/Moderate
  3. Moderate
  3.5- Moderate/Severe
Time Frame: Baseline, Week 16
Population: Subjects who completed week 16
Measure: Number; unit: Percent of participants
Arm/Group | Benzoyl Peroxide Wash -Clindamycin Foam | Benzoyl Peroxide Wash -Clindamycin Foam -Doxycycline Capsules
Number analyzed (Participants) | 10 | 12
Percent of participants
  % Clear skin | 0 | 8.3
  % Clear or Almost Clear | 0 | 8.3
  % Almost Clear | 30 | 25
  % Almost clear/ mild | 10 | 8.3
  % Mild | 10 | 25
  % Mild/ Moderate | 20 | 8.3
  % Moderate | 30 | 16.7

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Subjects who had visits at the first visit (Week 4) after baseline had AEs recorded.
Arm/Group | Benzoyl Peroxide Wash -Clindamycin Foam | Benzoyl Peroxide Wash -Clindamycin Foam -Doxycycline Capsules
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 4/13 | 4/14
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benzoyl Peroxide Wash -Clindamycin Foam (N=13) | Benzoyl Peroxide Wash -Clindamycin Foam -Doxycycline Capsules (N=14)
Stomach flu (Infections and infestations) | 1 (1) | 0 (0)
Cough (Infections and infestations) | 1 (1) | 0 (0)
Cold/ Cold symptoms (Infections and infestations) | 2 (3) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Fever (Infections and infestations) | 0 (0) | 1 (1)
Nausea/ vomiting (Infections and infestations) | 0 (0) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size did not provide adequate power. Even with the limited sample size, total lesion counts provides a more reliable view of the study data due to the greater number of lesions to work with.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days